CLINICAL TRIAL: NCT04563741
Title: MOVE!+UP: Testing a Tailored Weight Management Program for Veterans With PTSD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IIR 18-230; HX002755-01A2 (Other Grant/Funding Number: U.S. Department of Veterans Affairs)
Record Dates: First submitted 2020-09-08; First posted 2020-09-24 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: PTSD; Overweight; Obesity
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Overweight; Obesity

STUDY DESIGN:
Intervention Model Description: This is a hybrid type 1 trial with Veterans with PTSD who are classified as overweight or with obesity, and who are currently enrolled in PTSD care. Participants will be randomized to usual care enhanced with MOVE! (control) or usual care enhanced with MOVE!+UP (intervention).
Who Masked: Outcomes Assessor
Masking Description: Outcomes assessors will not know the treatment assignment. Because this is a behavioral intervention, with supervision provided by the lead investigator, the participants, care providers, and investigators will not be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- MOVE!+UP (intervention) (Experimental): usual care enhanced with MOVE!+UP (intervention)
  Interventions: Behavioral: MOVE!+UP
- MOVE! (control condition) (Active Comparator): usual care enhanced with MOVE! (control condition)
  Interventions: Behavioral: MOVE!

INTERVENTIONS:
Behavioral: MOVE!+UP — behavioral weight management intervention developed for Veterans with PTSD
  Arms: MOVE!+UP (intervention)
Behavioral: MOVE! — standard VA weight management intervention
  Arms: MOVE! (control condition)

SUMMARY:
Posttraumatic Stress Disorder (PTSD) is common among Veterans and results in poor psychological functioning, quality of life, and physical health. This includes having disproportionately high rates of obesity, in part due to PTSD symptoms interfering with physical activity and healthy diet. Unfortunately, Veterans with PTSD have poorer weight loss outcomes than those without PTSD in VA's existing weight management program, MOVE!. Based on pilot work, it appears that a weight management program that augments standard PTSD care and targets PTSD-related barriers to weight loss improves weight and PTSD symptoms. Whether it improves these issues more than standard VA care is in need of study, which is the focus of the proposed research. The proposed study also seeks to understand factors that would interfere with and facilitate implementing the program in VA if it is effective. This Veteran-centered, tailored weight loss program may efficiently benefit both physical and mental health of Veterans with PTSD, addressing standard care limitations.

DETAILED DESCRIPTION:
Background: Post-traumatic stress disorder (PTSD), prevalent among Veterans, puts Veterans at increased risk for obesity and related conditions. Veterans with PTSD lose less weight in VA's MOVE! weight management program, due to PTSD symptoms that interfere with activity and healthy diet. In addition, many Veterans who receive evidence-based PTSD treatment remain symptomatic. A behavioral weight loss program that augments standard PTSD care and targets PTSD-related weight loss barriers called MOVE!+UP was piloted and iteratively refined among 44 overweight Veterans with PTSD. The fully developed MOVE!+UP is led by a psychologist and a Veteran peer support counselor, who provide complementary expertise. It includes 16 group sessions with 90 minutes of general weight loss support, coupled with Cognitive Behavior Therapy skills to address PTSD-specific barriers. Each session also includes a 30-minute community walk to address hypervigilance-based activity barriers and enhance classroom-based learning. Veterans receive two individual dietician visits, and counseling calls as needed. The cohort receiving the final MOVE!+UP package reported high satisfaction and had better weight loss outcomes than Veterans with PTSD in the general MOVE! program. They also reported substantial PTSD symptom reduction. Treatment targets like eating behaviors, activity, and insomnia also improved. MOVE!+UP effectiveness must be tested in a randomized trial.

Significance/Impact: MOVE!+UP is timely and efficient, simultaneously addressing physical and mental health of a priority Veteran group. MOVE!+UP is positioned to address HSR&D priorities by promoting mental health and improving PTSD symptoms, access to care, and whole health. This study is aligned with HSR&D and ORD methodological priorities by using a hybrid type 1 trial. This study's cost and utilization analyses, and systematic identification of implementation barriers and facilitators, would place effectiveness findings in context and facilitate rapid translation to the field if MOVE!+UP is effective. This study will also provide insights about ways that general MOVE! and PTSD care can be enhanced to improve reach and effectiveness.

Innovation: MOVE!+UP is the first weight loss program designed to address obesity in Veterans with PTSD.

Specific Aims: This study proposes to enroll Veterans with PTSD who are classified as overweight or with obesity and who are engaged in PTSD care. They will be randomized to usual care enhanced with MOVE! (control) or usual care enhanced with MOVE!+UP (intervention), and is guided by three aims: 1) Test whether intervention participants have greater 6-month weight loss (primary outcome), and 6- and 12-month PTSD symptom reduction and 12-month weight loss (secondary exploratory outcomes), relative to controls; 2) Assess whether compared to control, intervention participants have greater improvements on 6-month treatment targets: physical activity, eating behavior, insomnia, depression, and social support; 3) Estimate intervention and control condition costs and utilization, and identify MOVE!+UP implementation barriers and facilitators, to contextualize Aim 1 and inform future implementation.

Methodology: Hybrid type 1 trial with 164 Veterans with PTSD who are classified as overweight or with obesity and are currently enrolled in PTSD care.

Implementation/Next Steps: This hybrid type 1 trial will provide data needed to prepare a MOVE!+UP implementation package for broader VA implementation if MOVE!+UP is effective. If it is not effective, Aims 2 and 3 will help understand how overweight Veterans with PTSD could be better supported in the future. Implementation activities would be coordinated with existing local, VISN, and national operational partners.

ELIGIBILITY:
Inclusion Criteria:

* PTSD Diagnosis: standard criteria for PTSD Checklist for DSM-5 (PCL-5): lifetime experience of trauma and a score of 33
* Overweight or obesity based on Body Mass Index (BMI) of 25 kg/m2
* Primary Care Provider or other physician approval
* Willing to participate in all intervention or control and assessment activities
* Enrolled in PTSD treatment
* Must have active VA Puget Sound Health Care System medical record.

Exclusion Criteria:

* Not fluent in English, severe hearing loss, no phone access
* Current MOVE! participation
* Current pregnancy
* Based on clinical judgment, would be unable to participate because of:

  * acutely exacerbated substance use, mental health, or chronic medical conditions
  * or moderate to severe chronic, progressive neurologic conditions such as Dementia
  * had bariatric surgery within the last 12 months or plan to undergo bariatric surgery within the next 6 months.
  * Report they cannot safely weigh themselves using the mailed study scale due to mobility issues or use of assistive devices
  * Baseline weight >440 lbs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 174 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2025-03-26 (Actual); Study Completion 2025-03-26 (Actual)

PRIMARY OUTCOMES:
weight (pounds) change | baseline and 6 months post-baseline
  This study's primary aims is to test whether intervention participants have greater 6-month weight loss, relative to controls.

SECONDARY OUTCOMES:
weight (pounds) | baseline and 12 months post-baseline
  Test whether intervention participants have greater long-term (12-month) weight loss, relative to controls.
PTSD symptom severity on the PTSD Checklist for DSM-5 | baseline and 6 and 12 months post-baseline
  Assess whether compared to control, intervention participants have greater improvements on 6- and 12-month PTSD symptom severity.

OTHER OUTCOMES:
insomnia measured with the Insomnia Severity Index | baseline and 6 months post-baseline
  Assess whether compared to control, intervention participants have greater improvements on 6-month insomnia severity.
average daily light, moderate, and vigorous physical activity measured with accelerometers | baseline and 6 months post-baseline
  Assess whether compared to control, intervention participants have greater improvements on 6-month accelerometry-based light, moderate, and vigorous physical activity.
Internalized weight bias measured with "Modified Weight Bias Internalization Scale" | baseline and 6 months post-baseline
  Assess whether compared to control, intervention participants have greater improvements on 6-month internalized weight bias.
depression severity measured with the Patient Health Questionnaire, 8-item version | baseline and 6 months post-baseline
  Assess whether compared to control, intervention participants have greater improvements on 6-month depression symptoms.
average daily moderate and vigorous physical activity measured with accelerometers | baseline and 6 months post-baseline
  Assess whether compared to control, intervention participants have greater improvements on 6-month accelerometry-based moderate and vigorous physical activity.
Eating habits measured with "PACE" eating habits measure | baseline and 6 months post-baseline
  Assess whether compared to control, intervention participants have greater improvements on 6-month eating habits
binge eating (yes vs. no) measured using an adapted Patient Health Questionnaire for DSM 5 criteria | baseline and 6 months post-baseline
  Assess whether compared to control, intervention participants have lower prevalence of engaging in binge eating at 6 months post-baseline.
night eating measured with the Night Eating Questionnaire | baseline and 6 months post-baseline
  Assess whether compared to control, intervention participants have greater improvements on 6-month night eating symptoms.
social support for physical activity and healthy eating measured with adapted Sallis measure | baseline and 6 months post-baseline
  Assess whether compared to control, intervention participants have greater improvements on 6-month social support for physical activity and healthy eating.
emotional eating measured with the Emotional Overeating Questionnaire | baseline and 6 months post-baseline
  Assess whether compared to control, intervention participants have greater improvements on 6-month emotional eating.
diet quality measured with "Starting the Conversation" | baseline and 6 months post-baseline
  Assess whether compared to control, intervention participants have greater improvements on 6-month diet quality.

CONTACTS AND LOCATIONS:
Overall Officials: Katherine D Hoerster, PhD MPH BA, Principal Investigator — VA Puget Sound Health Care System Seattle Division, Seattle, WA
Locations (1):
- VA Puget Sound Health Care System Seattle Division, Seattle, WA, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Hoerster KD, Tanksley L, Sulayman N, Bondzie J, Brier M, Damschroder L, Coggeshall S, Houseknecht D, Hunter-Merrill R, Monty G, Saelens BE, Sayre G, Simpson T, Wong E, Nelson K. Testing a tailored weight management program for veterans with PTSD: The MOVE! + UP randomized controlled trial. Contemp Clin Trials. 2021 Aug;107:106487. doi: 10.1016/j.cct.2021.106487. Epub 2021 Jun 16. PMID 34144246

DOCUMENTS (1):
  • Informed Consent Form (2023-10-13): https://cdn.clinicaltrials.gov/large-docs/41/NCT04563741/ICF_000.pdf